CLINICAL TRIAL: NCT00655252
Title: An Open-Label, Multi-Center, Expanded Access Study of RAD001 in Patients With Metastatic Carcinoma of the Kidney Who Are Intolerant of or Have Progressed Despite Any AvailableVascular Endothelial Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy
Brief Title: Expanded Access Study of RAD001 in Metastatic Renal Cell Cancer Patients Who Are Intolerant of or Who Have Failed Despite Prior Vascular Endothelial Growth Factor Therapy
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRAD001L2401
Record Dates: First submitted 2008-04-07; First posted 2008-04-09 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Metastatic Renal Cell Cancer
Keywords: Expanded access; metastatic renal cell cancer; progression despite VEGF receptors
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
This expanded access study is designed to provide RAD001 to patients with MRCC who are without satisfactory treatment alternatives, until RAD001 becomes commercially available.

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years old; metastatic renal cancer, intolerant of or failed sunitinib and/or sorafenib
* Adequate bone marrow function, liver function, renal function
* Adequate birth control

Exclusion criteria:

* Previously received RAD001 or other mTOR inhibitors, known hypersensitivity to rapamycin, chronic systemic treatment with corticosteroids or immunosuppressive agents (prednisone ≤ 20 mg/day for adrenal insufficiency OK
* Topical or inhaled steroids OK)
* Active bleeding
* Uncontrolled angina, CHF, heart attack ≤ 6 months, uncontrolled diabetes

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (84):
- United States (15):
  - Highlands oncology Group, PA, Springdale, Arkansas
  - University of Colorado Health Sciences Center/Anschutz Pavillion, Aurora, Colorado
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - MD Anderson Cancer Center - Orlando, Orlando, Florida
  - Indiana University Cancer center, Indianapolis, Indiana
  - The Cancer Institute, St. Joseph Medical Center, Towson, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Missouri Cancer Associates, Columbia, Missouri
  - Heartland Hematology-Oncology Associates, Inc., Kansas City, Missouri
  - Washington University/Siteman Cancer Center, St Louis, Missouri
  - Blumenthal Cancer Center/Carolinas Medical Center, Charlotte, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Cliveland Clinic Foundation, Cleveland, Ohio
  - Cleo Craig Memorial Cancer & Research Clinic, Lawton, Oklahoma
  - Cancer centers of the Carolinas, Greenville, South Carolina
- Novartis Investigative Site, Malvern, Australia
- Austria (4):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Brussels, Belgium
- Canada (8):
  - Moncton Hospital, Moncton, New Brunswick
  - QE ll Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Ontario
  - Lakeridhe Health Corp - Oshawa, Oshawa, Ontario
  - Sault Area Hospital - General Site, Sault Ste. Marie, Ontario
  - Les Urologues Associes du CHUM, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Germany (30):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bautzen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative site, Münster
  - Novartis Investidative Site, Nuremberg
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Wuppertal
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Beirut, Lebanon
- Norway (2):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Oslo
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Sankt Gallen
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (14):
  - Royal Bournemouth Hospital, Bournemouth
  - British Haematology and Oncology Centre, Bristol
  - Addenbrookes Hospital, Cambridge
  - CRUK, Glasgow
  - Southampton University Hospital NHS Trust,, Hampshire
  - Oncology & Haematology Clinical Tirals Unit, Leicester
  - Royal Free Hospital, London
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - Royal Marsden Hospital, London
  - The Christie Hospital, Manchester
  - Newcastle General Hospital, Newcastle
  - Mount Vernon Cancer Centre, Northwood
  - St Luke's Wing, Royal Surrey County Hospital, Surrey
  - Singleton Hospital, Swansea

REFERENCES:
- [Derived] Bracarda S, Rottey S, Bahl A, Eichelberg C, Mellado B, Mangel L, Cattaneo A, Panneerselvam A, Grunwald V. REACT expanded-access program in patients with metastatic renal cell carcinoma: real-world data from a European subanalysis. Future Oncol. 2015;11(21):2893-903. doi: 10.2217/fon.15.241. Epub 2015 Sep 17. PMID 26376939
- [Derived] Grunwald V, Karakiewicz PI, Bavbek SE, Miller K, Machiels JP, Lee SH, Larkin J, Bono P, Rha SY, Castellano D, Blank CU, Knox JJ, Hawkins R, Anak O, Rosamilia M, Booth J, Pirotta N, Bodrogi I; REACT Study Group. An international expanded-access programme of everolimus: addressing safety and efficacy in patients with metastatic renal cell carcinoma who progress after initial vascular endothelial growth factor receptor-tyrosine kinase inhibitor therapy. Eur J Cancer. 2012 Feb;48(3):324-32. doi: 10.1016/j.ejca.2011.06.054. Epub 2011 Jul 29. PMID 21803569
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com//webapp/etrials/DiseaseID97/Kidney-Cancer(renal-cell-cancer)-clinicaltrials.go